CLINICAL TRIAL: NCT07363148
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Clinical Trial to Investigate the Safety and Efficacy of MB-1 on Metabolic Health in Overweight and Obese Adults
Brief Title: A Clinical Trial to Investigate the Safety and Efficacy of MB-1 on Metabolic Health in Overweight and Obese Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arrae (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25ARCCM01
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Obese; Overweight Adults; Obese Adults; Body Weight Control; BMI
Keywords: Arrae; MB-1; Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MB-1 (Experimental): MB-1 contains African mango seed (Irvingia Gabonensis), Cissus leaf (Cissus quadrangularis) extract, Grains of Paradise (Aframomum melegueta), Bifidobacterium Lactis (B. lactis) B420, Green tea extract (standardized to 92 ± 2.5 % caffeine), Green tea extract (Camellia sinensis), Vitamin B6, and Chromium Picolinate.
  Interventions: Dietary Supplement: MB-1
- Placebo (Experimental): Placebo contains white rice flour
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: MB-1 — Participants will be instructed to take two capsules every morning with a meal for the duration of the study starting on Day 1.
  Arms: MB-1
Other: Placebo — Participants will be instructed to take two capsules every morning with a meal for the duration of the study starting on Day 1.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the safety and efficacy of MB-1 on metabolic health in overweight and obese adults. The main question it aims to answer is:

What is the difference in change in body weight and body mass index (BMI) from baseline at Day 84 between MB-1 and placebo?

Participants will be provided MB-1 or placebo and be assessed for anthropometric measurements, blood pressure, heart rate, and asked to complete appetite and satiety questionnaires and undergo a DEXA scan.

ELIGIBILITY:
Inclusion Criteria:

1. Males & females aged 18-65 years, inclusive
2. BMI of 25.0 to ≤ 34.9 kg/m²
3. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically-approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle and agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence and agrees to use contraception if planning on becoming sexually active during the study
4. Stable body weight defined as a <5% change in body weight in the three months prior to baseline as assessed by the QI
5. Abdominal obesity: Waist circumference of > 94 cm (37 inches) in men and > 80 cm (31.5 inches) in women
6. Willingness to complete questionnaires, records and diaries associated with the study and to complete all clinic visits
7. Agrees to maintain current lifestyle habits (diet, medications, supplements, and sleep) as much as possible throughout the study
8. Provided voluntary, written, informed consent to participate in the study
9. Healthy as determined by medical history as assessed by Qualified Investigator (QI)

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, or intolerance preventing consumption of the investigational product or placebo ingredients
3. Gastric bypass surgery or other surgeries to induce weight loss
4. Metal implants or other physical characteristics/limitations that may affect DEXA scan results as assessed by the QI
5. Currently taking weight loss medications or participated in a weight loss program within the past three months as assessed by the QI
6. Current or history of eating disorders as assessed by the QI
7. Unstable metabolic disease or chronic diseases as assessed by the QI
8. Current or history of any significant diseases of the gastrointestinal tract as assessed by the QI
9. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
10. Participants residing in the same household as another study participant unless they are enrolled consecutively (e.g. not actively enrolled at the same time)
11. Type I diabetes
12. Type II diabetes with HbA1c of ≥ 6.5% and/or if < 6 months of stable medication use
13. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
14. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
15. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
16. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
17. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
18. Individuals with an autoimmune disease or are immune compromised as assessed by the QI
19. Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis as assessed by the QI
20. Self-reported confirmation of blood/bleeding disorders as assessed by the QI
21. Chronic use of cannabinoid products (>2 times/week) as assessed by the QI. Occasional users will be required to washout and abstain for the duration of the study period
22. Regular use of tobacco or nicotine products in the past six months, as assessed by the QI. Occasional users will be required to washout and abstain for the duration of the study period
23. Alcohol intake average of >2 standard drinks per day as assessed by the QI
24. Alcohol or drug abuse within the last 12 months
25. Current use of prescribed and/or over-the-counter (OTC) medications, supplements, and/or consumption of food/drinks that may impact the efficacy and/or safety of the investigational product (Section 7.3)
26. Blood donation 30 days prior to baseline, during the study, or a planned donation within 30 days of the last study visit
27. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
28. Individuals who are unable to give informed consent
29. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The difference in change in body weight and body mass index (BMI) between MB-1 and placebo | Day 0 to 84
  The difference in change in body weight and body mass index (BMI) from baseline at Day 84 between MB-1 and placebo

SECONDARY OUTCOMES:
The difference in change in body weight and BMI between MB-1 and placebo | Day 0 to 42
  The difference in change in body weight and BMI from baseline at Day 42 between MB-1 and placebo
The difference in change in anthropometric measures (waist, arm, thigh, and hip circumference) between MB-1 and placebo | Day 0 to 42
  The difference in change in anthropometric measures (waist, arm, thigh, and hip circumference) from baseline at Days 42 between MB-1 and placebo
The difference in change in anthropometric measures (waist, arm, thigh, and hip circumference) between MB-1 and placebo | Day 0 to 84
  The difference in change in anthropometric measures (waist, arm, thigh, and hip circumference) from baseline at Day 84 between MB-1 and placebo
The difference in change in body composition (fat and muscle mass) between MB-1 and placebo as assessed by Dual-Energy X-Ray Absorption (DEXA) | Day 0 to 84
  The difference in change in body composition (fat and muscle mass) from baseline at Day 84 between MB-1 and placebo as assessed by Dual-Energy X-Ray Absorption (DEXA)
The difference in change in Resting Energy Expenditure (REE), adjusted for bodyweight and body composition between MB-1 and placebo | Day 0 to 84
  The difference in change in Resting Energy Expenditure (REE), adjusted for bodyweight and body composition from baseline at Day 84 between MB-1 and placebo
The difference in change in glycemic markers between MB-1 and placebo as assessed by fasting blood glucose | Day 0 to 84
  The difference in change in glycemic markers from baseline at Day 84 between MB-1 and placebo as assessed by fasting blood glucose
The difference in change in glycemic markers between MB-1 and placebo as assessed by Glycated hemoglobin (HbA1c) | Day 0 to 84
  The difference in change in glycemic markers from baseline at Day 84 between MB-1 and placebo as assessed by Glycated hemoglobin (HbA1c)
The difference in change in lipid profile between MB-1 and placebo | Day 0 to 84
  The difference in change in lipid profile: total cholesterol (TC) between MB-1 and placebo
The difference in change in lipid profile between MB-1 and placebo | Day 0 to 84
  The difference in change in lipid profile: low-density lipoprotein cholesterol (LDL-C between MB-1 and placebo
The difference in change in lipid profile between MB-1 and placebo | Day 0 to 84
  The difference in change in lipid profile: high-density lipoprotein cholesterol (HDL-C) between MB-1 and placebo
The difference in change in lipid profile between MB-1 and placebo | Day 0 to 84
  The difference in change in lipid profile: non-HDL-C between MB-1 and placebo
The difference in change in lipid profile between MB-1 and placebo | Day 0 to 84
  The difference in change in lipid profile: triglycerides (TG) between MB-1 and placebo
The difference in change in lipid profile between MB-1 and placebo | Day 0 to 84
  The difference in change in lipid profile: TG/HDL-C, TC/HDL-C and LDL-C/HDL-C between MB-1 and placebo
The difference in change in leptin and adiponectin between MB-1 and placebo | Day 0 to 84
  The difference in change in leptin and adiponectin from baseline at Day 84 between MB-1 and placebo
The difference in change in ratings of appetite and satiety between MB-1 and placebo as assessed by the weekly Appetite and Satiety Likert scales. | Day 0 to 84
  The difference in change in ratings of appetite and satiety from baseline at Day 84 between MB-1 and placebo as assessed by the weekly Appetite and Satiety Likert scales. On a scale of 0 to 10, with 0 being "I was not hungry at all" and 10 being "I have never been more hungry"
The difference in change in ratings of energy and cravings between MB-1 and placebo as assessed by the weekly Appetite and Satiety Likert scales. | Day 0 to 84
  The difference in change in ratings of energy and cravings from baseline at Day 84 between MB-1 and placebo as assessed by the weekly Energy and Cravings Likert scales. On a scale of 0 to 10, with 0 being "I had no energy" and 10 being "I have never had more energy"

OTHER OUTCOMES:
Incidence of post-emergent adverse events (AE) | Day 0 to 84
  Incidence of post-emergent adverse events (AE)
Clinically relevant changes in heart rate (HR) after supplementation | Day 0 to 84
  Clinically relevant changes in heart rate (HR) after supplementation
Clinically relevant changes in blood pressure (BP) after supplementation | Day 0 to 84
  Clinically relevant changes in blood pressure (BP) after supplementation

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada